CLINICAL TRIAL: NCT01881841
Title: Computer Adaptation of Screening, Brief MET Intervention to Reduce Teen Drinking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Sion Kim Harris, Assistant Professor of Pediatrics, Harvard Medical School; Co-Director, Center for Adolescent Substance Abuse Research, Boston Children's Hospital, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JRKnightR34PA-13-078
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Alcohol Abuse; Tobacco Use Disorder; Substance Use
Keywords: Alcohol abuse; Substance use; Tobacco use disorder; Motivational Enhancement Therapy; Adolescents
MeSH Terms: conditions — Alcoholism; Tobacco Use Disorder; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment As Usual (No Intervention): Those randomized to Treatment as Usual (TAU) will not complete cMET but will receive standard treatment from the doctor.
- cMET (Experimental): Those randomized to cMET will complete a 2-session computerized Motivational Enhancement Therapy (cMET) intervention.
  Interventions: Behavioral: cMET

INTERVENTIONS:
Behavioral: cMET — Those in cMET complete the 2-session self-administered computerized intervention which includes 8 exercises designed to encourage adolescents to evaluate the impact of alcohol and other substance use on their health and well-being and consider changing their use.
  Other Names: Computerized Motivational Enhancement Therapy intervention
  Arms: cMET

SUMMARY:
The goal of this project is to evaluate the feasibility, acceptability, and effect size of a new computerized Motivational Enhancement Therapy (cMET) intervention for alcohol-involved adolescents in primary care.

DETAILED DESCRIPTION:
The study aims are to:

1. Assess cMET feasibility and acceptability and estimate its effect size on underage drinking. Hypothesis: Among 14- to 20-yr-old primary care patients, those receiving cMET will have lower rates of any alcohol use, days of alcohol use, drinks per drinking day, and days of heavy episodic drinking, than those receiving treatment as usual.
2. Estimate effect sizes for tobacco, cannabis, and other drug use, and other substance-related risks and outcomes including substance-related driving/riding, and experience of substance-related problems.
3. Identify potential moderators and mediators of cMET's effect.

ELIGIBILITY:
Inclusion Criteria:

* 14- to 20- yr-olds
* arriving for routine care to one of our participating pediatric practices (Lexington Pediatrics, Lexington, MA; East Boston Community Health Center, Longwood Pediatrics, Tufts Medical Center Adolescent Clinic, Boston, MA; Cambridge Health Alliance Dept. of Pediatrics, Cambridge, MA)
* any alcohol use days in the past 90 days,
* have an email address and internet access at home, school, or library
* provide informed assent/consent.

Exclusion Criteria:

* unable to read or understand English,
* living away at college at the time of the recruitment visit,
* not available for computer/telephone follow-ups,
* judged by the provider to be medically or emotionally unstable at the time of the visit.

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Alcohol use | up to 9-months follow-up
  The study investigators will measure the past 90 day alcohol use at 3-, 6-, and 9-months follow-up.

SECONDARY OUTCOMES:
Drinks per drinking day | up to 9-months follow-up
  The study investigators will measure the number of drinks per drinking day in the past 90 days at 3-, 6-, and 9-months follow-up

OTHER OUTCOMES:
Heavy episodic drinking | up to 9-months follow-up
  The study investigators will measure the occurrences of heavy episodic drinking in the past 90 days at 3-, 6-, and 9-months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: John R Knight, MD, Principal Investigator — Boston Children's Hospital; Sion K Harris, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web site of the Center for Adolescent Substance Abuse Research at Boston Children's Hospital — http://www.ceasar.org